CLINICAL TRIAL: NCT00816582
Title: A Phase II Clinical Trial to Evaluate 18F-Fluoroestradiol Positron Emission Tomography / Computerized Tomography (PET/CT) Guided Fulvestrant Therapy for Patients With Recurrent or Metastatic Breast Cancer
Brief Title: PET/CT Guided Fulvestrant Therapy for Patients With Recurrent or Metastatic Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PET/CT Breast
Record Dates: First submitted 2008-12-30; First posted 2009-01-01 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Post-menopausal hormone receptor positive recurrent/metastatic breast cancer.; PET/CT; Recurrent or metastatic
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET/CT Guided FES Therapy (Experimental): All subjects will be seen at baseline and then monthly until month 6 of fulvestrant therapy unless clinical or radiological progression or unacceptable toxicity earlier than month 6.
  Interventions: Procedure: Diagnostic Imaging: 18F-FDG PET/CT Scan - Baseline; Procedure: Diagnostic Imaging: 18F-FES PET/CT - Baseline; Procedure: Diagnostic Imaging: 18F-FES PET/CT - 3 month follow-up

INTERVENTIONS:
Procedure: Diagnostic Imaging: 18F-FDG PET/CT Scan - Baseline — A18F-FDG PET/CT scan performed at baseline, prior to starting the fulvestrant treatment, to identify the sites involved by the subject's cancer.
Procedure: Diagnostic Imaging: 18F-FES PET/CT - Baseline — A 18F-FES PET/CT scan performed at baseline, prior to starting the fulvestrant treatment, to determine the hormone receptor content of the sites involved by the breast cancer.
Procedure: Diagnostic Imaging: 18F-FES PET/CT - 3 month follow-up — A 18F-FES PET/CT scan performed after three (3) monthly injections of fulvestrant to determine whether estrogen uptake is blocked by fulvestrant.

SUMMARY:
Purpose:

To determine whether [18F]FES can predict clinical benefit (defined as complete response, partial response and stable disease ≥ 6 months) to fulvestrant (250 mg IM q 28 days) in post-menopausal women with recurrent or metastatic ER+ breast cancer who are candidates for further hormonal therapy.

DETAILED DESCRIPTION:
The majority of women diagnosed with breast cancer are post-menopausal, of which up to 75% are estrogen (ER) and/or progesterone receptor (PR) positive. Even in pre-menopausal breast cancer over half of all patients will have expression of these hormone receptors. Thus therapeutic strategies targeting the estrogen receptor or its ligand are the most common treatment offered in breast cancer. Despite substantial benefits now demonstrated with selective estrogen receptor modulators (e.g. tamoxifen) and aromatase inhibitors (e.g. anastrazole, letrozole and exemestane), a significant proportion of patients will still unfortunately have or develop resistance to these hormonal therapies.

Despite approximately two-thirds of patients who are prescribed fulvestrant following prior hormonal agents not benefiting from this therapy, clinicians are still offering this option to all suitable women because of the lack of a better means of identifying the individual responders.

To assess whether the recommended treatment is beneficial to a specific individual, the disease burden is assessed before and following treatment. Conventional imaging techniques such as the bone scan or computerized tomography (CT) can take several months to show a successful response to treatment. Positron emission tomography (PET) can improve the evaluation of women with breast cancer by providing an accurate assessment of the extent of disease and unique information about tumor biology such as metabolic activity.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal (≥ 60 years old, or age ≥ 45 years with amenorrhea for > 12 months or follicle stimulating hormone and estrogen levels within post-menopausal range, or prior bilateral oophorectomy)
* hormone receptor positive (ER and/or PgR) disease as determined locally
* WHO performance status 0-2
* life expectancy of ≥ 3 months
* the presence of at least one measurable or evaluable (non-measurable) lesion
* informed consent prior to any study procedures

Exclusion Criteria:

* life threatening metastatic visceral disease
* brain or leptomeningeal metastases
* prior exposure to fulvestrant
* history of bleeding diathesis or need for long term anti-coagulation

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2014-09-17 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | 24 weeks
  CBR is defined as a patient having a best overall response of a complete response (CR), partial response (PR), or stable disease for at least 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chia, MD, Principal Investigator — BC Cancer Agency - Vancouver Centre
Locations (4):
- Canada (4):
  - BC Cancer Agency - Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency - Fraser Valley, Surrey, British Columbia
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver Island, Victoria, British Columbia